CLINICAL TRIAL: NCT01942421
Title: Ocular Surface Reconstruction With Cultivated Autologus Mucosal Epithelial Transplantation.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pinnita Prabhasawat, Associate professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 639/2551(EC2)
Record Dates: First submitted 2011-12-06; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Ocular Surface Disease
Keywords: Limbal deficiency; Cultivated limbal transplantation; Ex vivo limbal transplantation; Cultivated autologous mucosal epithelial transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cultivated mucosal epithelial transplant (Experimental): Cultivated mucosal epithelial transplantaion to limbal deficiency patients
  Interventions: Procedure: Cultivated mucosal epithelial transplantation

INTERVENTIONS:
Procedure: Cultivated mucosal epithelial transplantation — cultivated autologous mucosal epithelium, then transplant to limbal stem cell deficiency patients.

SUMMARY:
The purpose of this study is to elucidate the appropriate condition of developing cultivated autologous oral mucosal epithelial graft and evaluate the surgical outcome of transplantation of the cultivated cells in the patients.

DETAILED DESCRIPTION:
Ocular surface damage caused by severe ocular surface diseases. Corneal limbal stem cell transplantation has been demonstrated to improve the outcome of ocular surface reconstruction. However, the conventional management of allograft limbal transplantation generally has unsatisfactory outcome because of high risk of rejection and requires long-life immunosuppressive medications. Ocular surface reconstruction with cultivated autologous mucosal epithelial transplantation is served to improve the surgical results of ocular surface reconstruction and decrease the use of immunosuppressive medications

ELIGIBILITY:
Inclusion Criteria:

* Bilateral limbal stem cell deficiency proved by specific clinical features and impression cytology

Exclusion Criteria:

* Age under 18
* Active ocular infection, Severe dry eye, Uncontrolled glaucoma
* Immunocompromised host
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Ocular surface clinical and pathological status(signs of limbal deficiency and immunopathological markers)after the surgery | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Pinnita Prabhasawat, MD, Principal Investigator — Mahidol University
Locations (1):
- Pinnita Prabhasawat, MD, Bangkok, Thailand, Thailand